CLINICAL TRIAL: NCT03784235
Title: Study of Subchondral Bone Remodeling With 18F NaF-PET / CT in Patients With Patellofemoral Pain. A Substudy for: Comparative Effectiveness of Therapeutic Hip and Knee Exercise for Patellofemoral Pain: a Pragmatic Randomised Trial (the COMPETE Trial)
Brief Title: Bone Metabolic Activity in the Patellofemoral Joint in Patients With Unilateral PFP
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Rudi Neergaard Hansen, PT, MSc., University Hospital Bispebjerg and Frederiksberg
Other Study IDs: BFH_NaF-PET
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 18F NaF-PET/CT and cone beam CT scans — Cross sectional measures of 18F NaF-PET/CT and cone beam CT scans

SUMMARY:
This study aims to examine whether individuals with unilateral patellofemoral pain (PFP) have increased subchondral bone remodelling and thus increased 18F Sodium Fluoride (18F-NaF) uptake in the painful knee compared to the opposite knee measured by simultaneous positron emission tomography and computed tomography (PET/CT) and to examine whether the increased uptake is associated with pain intensity, with patient-reported function and with pain localization. Furthermore we aim to investigate the effect of an acute patellofemoral loading bout on the bone remodelling.

DETAILED DESCRIPTION:
Patellofemoral pain (PFP) is a highly prevalent musculoskeletal condition mainly affecting younger people, causing pain, physical disability, and reduced quality of life. The cause of PFP is still unknown. It is, i.e., unclear whether there is a link between PFP and changes in the cartilaginous (subchondral) bone in the joint between the patella and the femur.

Our goals are to use 18F NaF PET/CT to evaluate whether subjects with unilateral patellofemoral pain exhibit elevated bone metabolic activity in the painful knee compared to the pain free knee and to determine whether bone metabolic activity correlates with pain intensity and location of pain. Furthermore, we aim to investigate the effects of acute loading on the bone metabolic activity.

The primary objective of this cross-sectional study is to assess whether patients with unilateral PFP have increased bone metabolic activity in the painful knee compared to the pain free knee. We will assess quantitative parameters indicative of bone metabolic activity (Standardized Uptake Value (SUV) and kinetic data) and compare values between the painful knee and the pain free knee. The secondary objectives are to 1) determine whether a bout of single leg weight bearing knee bends standing on a wedge result in increased bone metabolic activity acutely in the painful knee compared to the pain free knee, and 2) identify "hot" regions of abnormal tracer uptake and compare area and SUV values between the painful knee and the pain free knee.

An explorative objective is to determine the correlation between bone metabolic activity and pain intensity and location of pain.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of PFP in at least one knee confirmed by an experienced sports medicine doctor.
* Visual analogue score rating of pain during activities of daily living during the previous week at a minimum of 3 on a 10 cm scale.
* Insidious onset of symptoms unrelated to trauma and persistent for at least 4 weeks.
* Pain in the anterior knee associated with at least 3 of the following:

  * During or after activity
  * Prolonged sitting
  * Stair ascent or descent
  * Squatting

Exclusion Criteria:

* Meniscal or other intra-articular injury
* Cruciate or collateral ligament laxity or tenderness
* Patellar tendon, iliotibial band, or pes anserine tenderness
* Osgood-Schlatter or Sinding-Larsen-Johansson syndrome
* History of recurrent patellar subluxation or dislocation
* History of surgery to the knee joint
* History of head injury or vestibular disorder within the last 6 months
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (n = 30) with unilateral anterior knee pain / PFP (3> 10 NRS) will be included from the main study.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
18F NaF-PET/CT uptake | Cross sectional assessment at baseline, i.e., before the loading programme.
  Difference between painful knee and contralateral knee in mean, peak and maximum Standardized Uptake Value (SUV) and in kinetic parameters

SECONDARY OUTCOMES:
18F NaF-PET/CT uptake | Assessed before and after an acute loading programme (on the same day).
  Response to acute patellofemoral joint loading in mean, peak and maximum SUV and in kinetic parameters. The outcome represents changes in the parameters from before to after the loading programme
Regions of abnormal tracer uptake | Cross sectional assessment at baseline, i.e., before the loading programme
  Identify "hot" regions of abnormal tracer uptake and compare area and SUV values between the painful knee and the pain free knee

OTHER OUTCOMES:
18F NaF-PET/CT uptake and pain intensity, pain localization and physical function. | Cross sectional assessment at baseline, i.e., before the loading programme
  Correlation between tracer uptake parameters and pain intensity measured by pain algometry, pain localization measured by pain drawings and physical function measured by the Anterior Knee Pain Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, København NV, Denmark

IPD SHARING:
Plan to Share IPD: No